CLINICAL TRIAL: NCT06939595
Title: A Double-Blind, Randomized, Active-Controlled, Parallel-Group, Phase 3 Study to Compare Efficacy and Safety of CT-P51 and Keytruda in Combination With Platinum-Pemetrexed Chemotherapy in Patients With Previously Untreated Metastatic Non-Squamous Non-Small Cell Lung Cancer
Brief Title: A Study to Compare Effects and Safety of CT-P51 and Keytruda in Patients With Previously Untreated Metastatic Lung Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-P51 3.1
Record Dates: First submitted 2025-04-21; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Non Squamous Non Small Cell Lung Cancer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CT-P51 (Experimental)
  Interventions: Drug: CT-P51
- EU-approved Keytruda (Active Comparator)
  Interventions: Drug: EU-approved Keytruda

INTERVENTIONS:
Drug: CT-P51 — CT-P51 200mg with pemetrexed and cisplatin or carboplatin will be administered every 3 weeks for a maximum of 4 cycles followed by CT-P51 or Keytruda and pemetrexed every 3 weeks
  Arms: CT-P51
Drug: EU-approved Keytruda — Keytruda 200mg with pemetrexed and cisplatin or carboplatin will be administered every 3 weeks for a maximum of 4 cycles followed by CT-P51 or Keytruda and pemetrexed every 3 weeks
  Arms: EU-approved Keytruda

SUMMARY:
The goal of this Phase 3 clinical trial is to compare efficacy and safety of CT-P51 and European Union (EU) approved Keytruda in combination with platinum pemetrexed chemotherapy in patients with previously untreated metastatic nsNSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Stage IV, non squamous NSCLC
* Have not received any prior systemic anti-cancer therapy for metastatic NSCLC
* Have at least 1 measurable lesion per RECIST version 1.1

Exclusion Criteria:

* Have predominantly squamous cell histology NSCLC.
* Hypersensitivity or contraindication to any component of the study drug, pemetrexed and cisplatin or carboplatin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 606 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
ORR based on the confirmed best overall response (BOR) by the end of Cycle 11 according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 | Up to 34 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- ltd "Institute of Clinical Oncology", Tbilisi, Georgia